CLINICAL TRIAL: NCT05477914
Title: Assesment of Knowledge,Attitude and Practice of Pregnant Women Regarding Iron,Folic Acid and Multivitamins at AlMonshah District.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Somia Saadeldin Abdelhafez, resident doctor at family medicine department at almonshah health administration, Sohag University
Other Study IDs: Soh-Med-22-07-03
Record Dates: First submitted 2022-07-19; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnare about nutritional knowledge of pregnant women

SUMMARY:
Anaemia is defined as the lack of functioning red blood cells (RBCs) that leads to a decrease in the ability to carry oxygen causing a lot of complications during life time.

Iron deficiency anaemia is a main public health problem in all countries. Over 30% of the world's population had anaemia; 4.3%-20% and 30%-48% respectively in developed and developing countries are affected by iron deficiency anaemia. Globally, it is estimated that roughly 38% of pregnant females, 29% non-pregnant women, and 29% of all females of reproductive age are diagnosed to have anaemia .

WHO suggested a standard daily dose of 30 to 60 mg of iron and 400 µg of folic acid supplements to prevent anaemia in pregnancy. This dose of iron and folic acid should be taken ideally before gestation with the earliest possible time and must be continued throughout the gestational period.

During pregnancy it is important to take adequate nutrition which is essential for optimal growth of the foetus and decrease in the incidence of congenital anomalies. adequate dietary intake of proteins and energy is not enough for normal weight of the new-born, decrease in vitamins and minerals can adversely affect the weight of the new- born .

The prevalence of neural tube defects, low-birth weights, small babies for gestational age and maternal anaemia can be reduced by adequate intake of iron and folic acid supplements during pregnancy. A lot of studies show the same positive results for the intake of multivitamins ,but iron and folic acid are the most important .

A lot of studies show the importance of the relationship between iron and folic acid supplement or multivitamins intake and the socio-economic factors as age, level of education, residence, marital status, parity, economic status, prenatal circumstances. There are association between more intake of supplements during pregnancy and a higher socioeconomic levels , level of education and use of prenatal medical services in studies conducted in Finland . The detection of anaemia in pregnancy is based on the examination of haemoglobin (Hb) levels at the first antenatal care visit.

If the haemoglobin level is <11.9%, the pregnant woman is declared anaemic and should be given supplements of 60 mg iron tablets and 0.5 mg folic acid. This supplement is taken regularly 1 tablet per day for 90 consecutive days. If the haemoglobin level is still <11.9%, then the administration of iron tablets is continued. However, in practice, not all pregnant women take tablets regularly. This could be due to inadequate knowledge about the importance of iron tablets for pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who are resident in Almonshah district, Sohag and attend the mentioned health centers for antenatal care services.

Exclusion Criteria:

* 1- Women who refuse to participate in the study. 2- Presence of pregnancy complications. 3- Presence of psychiatric or cognitive diseases

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — females
Study Population: All pregnant women who are resident in Almonshah district, Sohag and attend the mentioned health centers for antenatal care services
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge,Attitude and Practice of Pregnant Women Regarding Iron,Folic Acid and Multivitamins | 1 month after recruitment of the participants
  using standradized questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Popa AD, Nita O, Graur Arhire LI, Popescu RM, Botnariu GE, Mihalache L, Graur M. Nutritional knowledge as a determinant of vitamin and mineral supplementation during pregnancy. BMC Public Health. 2013 Dec 1;13:1105. doi: 10.1186/1471-2458-13-1105. PMID 24289203
- [Background] Arkkola T, Uusitalo U, Pietikainen M, Metsala J, Kronberg-Kippila C, Erkkola M, Veijola R, Knip M, Virtanen SM, Ovaskainen ML. Dietary intake and use of dietary supplements in relation to demographic variables among pregnant Finnish women. Br J Nutr. 2006 Nov;96(5):913-20. doi: 10.1017/bjn20061929. PMID 17092382